CLINICAL TRIAL: NCT02920190
Title: Reduction of Antigen-Lipid-Driven Monoclonal Gammopathies by Targeting Epicardial Fat and Its Lipids Content With Liraglutide: A Glucagon Like Peptide-1 Receptor Analogue (GLP-1RA)
Brief Title: Antigen-Lipid-Driven Monoclonal Gammopathies Targeting Epicardial Fat
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funds to cover the costs of the study medications
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, James Hoffman, MD, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20160568
Record Dates: First submitted 2016-08-22; First posted 2016-09-30 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Monoclonal Gammopathies; Overweight; Obesity
MeSH Terms: conditions — Paraproteinemias; Overweight; Obesity | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Liraglutide Group (Experimental): Participants in this group will receive the Liraglutide intervention for 12 months
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — 1.8 mg Liraglutide administered subcutaneously once daily for 12 consecutive months
  Other Names: Victoza

SUMMARY:
The purpose of this research study is to learn about the effect of Liraglutide (Victoza) on the fat of the heart and some fat cells in blood.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥27 kg/m2
* At least one overweight/obesity related comorbidity (such as type 2 diabetes, pre-diabetes [IFG, IGT], hypertension, dyslipidemia)
* Age > 18 and < 70 years old

Exclusion Criteria:

* Known contra-indications to Liraglutide, such as previous history of pancreatitis or medullary thyroid carcinoma, personal or family history of MEN, in accordance with risks and safety information included in the latest updated Prescribing Information for Victoza®
* Type 1 diabetes, as defined by American Diabetes Association (ADA) criteria
* Insulin dependent or treated type 2 diabetes
* Current use of other injectable incretins
* History of diabetes ketoacidosis
* Advanced Chronic Kidney Disease, as defined by Glomerular Filtration Rate (GFR) < 30 mL/min/1.73m2
* Clinical signs or symptoms of New York Heart Association (NYHA) class III-IV heart failure
* Clinical or laboratory evidences of chronic active liver diseases
* Acute or chronic infective diseases
* Known or suspected allergy to Liraglutide, excipients, or related products
* Pregnant, breast-feeding or the intention of becoming pregnant
* Females of childbearing potential who are not using adequate contraceptive methods

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Epicardial Fat Thickness | Baseline, 12 months
  Epicardial fat thickness measured in mm via ultrasound

SECONDARY OUTCOMES:
Change in serum immunoglobulins | Baseline, 12 months
  Immunoglobin levels assessed in g/L will be evaluated using serum blood samples
Change in plasma ceramide levels | Baseline, 12 months
  Plasma ceramide levels will be evaluated in umol/L

CONTACTS AND LOCATIONS:
Overall Officials: James Hoffman, MD, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: No